CLINICAL TRIAL: NCT04951921
Title: Precision Medicine Imaging for Cervical Cancer: Integrating MR Fingerprinting, Dynamic Nuclear Polarization (DNP)-MRI and Artificial Intelligence Radiomics
Brief Title: Hyperpolarized 13C Pyruvate MRI for Early Immune Evaluation in Cervical Cancer Patients At Baseline and CCRT Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Gigin Lin, Clinical Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201702080A0
Record Dates: First submitted 2021-06-21; First posted 2021-07-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
Keywords: Hyperpolarized 13C pyruvate; Dynamic nuclear polarization; Artificial intelligence; Cervical cancer; Magnetic resonance fingerprinting; Precision medicine; Radiomics
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hyperpolarized 13C pyruvate DNP-MRI scan (Experimental): Patients receive hyperpolarized 13C pyruvate through IV injection less than 1-2 minute then undergo MRI over 3-5 minutes at baseline and 2 weeks after CCRT treatment. Total 2 times of MRI scan.
  Interventions: Drug: Hyperpolarized 13C Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13C Pyruvate — Procedure: Magnetic Resonance Imaging Undergo 1H-MRI of DWI/MRF/CEST for tumor cite following by 13C DNP-MRI for spleen for 3-5 minutes after hyperpolarized 13C pyruvate injection
  Other Names: Hyperpolarized Carbon C 13 Pyruvate; Hyperpolarized Pyruvate (13C)

SUMMARY:
In this single armed, single-center, case-controlled study, the investigators will conduct a prospective trial and integrate the most advanced imaging technology to medical practice, attempting to solve the problem detected by radiomics approach. The investigators plan a 3-year project with non-randomized, single group assignment observational study design. Thirty participants with diagnosed LACC that are to receive CCRT are to be recruited for this prospective single institutional study from Chang Gung Memorial Hospital at Linkou (CGMH). Standard-of-care MRI/CT that is required for staging will be the first line screening method. A tumor biopsy and routine blood test will be obtained at the time of the initial clinic visit. Participants eligible for this study will receive two investigative exams-MRF, CEST, DNP-MRI MRI and Metabolomics, at baseline and the 2-week during CCRT.

The new imaging methods being tested are MRF and CEST without contrast enhancement, and DNP-MRI which provides quantitative measurement of the metabolism occurring within cancer cells. It also involves injection of a contrast agent-Hyperpolarized pyruvate (13C) Injection. The participants will be injected with the study drug at a dose of 0.43 ml/kg and then receive MRI scan.

DETAILED DESCRIPTION:
Primary objective

1. Bridging the Gap between Imaging and Biology. DNP is the only technology that can measure real-time flux of pyruvate to lactate conversion and mitochondria metabolism. DNP-MRI will combine the strength of MRI (anatomy, tissue contrast via MRF, CEST and DWI) and DNP (biochemistry measurement), and the blood/urine metabolomics approach, to noninvasively bring more insightful information for clinical application.
2. Precision Medicine for Precision Response Prediction. Although AI or deep learning can identify high-risk patient for particularly treatment (CCRT in this project), the predictive model is based on prior database rather than this particular patient. The investigators urgently need a non-invasive precise measurement to monitor the response in a real-world situation, to reduce the treatment uncertainty, to select the most cost-effective treatment. This is of paramount importance for the more advanced treatment i.e. target therapy, immunotherapy etc. The investigators did not intend to change the standard-of-care but the information provided by this study will help to investigate the fundamental mechanisms hence providing hopes for alternative treatments.
3. Infrastructures for MR Fingerprinting and Dynamic Nuclear Polarization (DNP)-MRI Research for Taiwanese researchers. The investigators are very grateful to be able to install the first DNP system dedicated to human research in Asia and would like to introduce this novel technology to Taiwan. Currently, human DNP study has only been conducted in the USA (UCSF, MD Anderson Cancer Center and Memorial Sloan-Kettering Cancer Center) and the UK (University College of London, Oxford and Cambridge) and Canada (Toronto University). Based on our preliminary efforts of tracer preparation, multi-nuclei scanning equipment and dedicated pulse sequences, the investigators aim to build infrastructures for MR Fingerprinting and DNP-MRI Research for Taiwanese research groups.

Secondary objective

1. Translate technical advancements to clinically applicable tools
2. Converge integrated information to construct the prediction model
3. Establish the delta radiomics prediction model with biological meaningfulness

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed carcinoma of the uterine cervix.
2. Age ≥ 20 years.
3. Clinical International Federation of Gynecology and Obstetrics (FIGO) stage IB2-IV.
4. Tumor diameter ≥ 4 cm, verified by MRI or CT.
5. Scheduled curative-intent non-surgical treatment.

Exclusion Criteria:

1. Contraindication to MRI study (e.g. claustrophobia, cardiac pacemaker, metal implants in pelvis).
2. Inadequate marrow, liver and renal functions.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Pregnant or breast-feeding women.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
MRI size measurement of the primary tumor | Change from baseline in tumor size at 3 months
  Tumor size measurement by regular MRI

SECONDARY OUTCOMES:
Recurrent rate | Follow-up for 5 years
  Follow-up recurrent rate

CONTACTS AND LOCATIONS:
Overall Officials: Gigin Lin, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Guishan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin G, Hsieh CY, Lai YC, Wang CC, Lin Y, Lu KY, Chai WY, Chen AP, Yen TC, Ng SH, Lai CH. Hyperpolarized [1-13C]-pyruvate MRS evaluates immune potential and predicts response to radiotherapy in cervical cancer. Eur Radiol Exp. 2024 Apr 10;8(1):46. doi: 10.1186/s41747-024-00445-1. PMID 38594558